CLINICAL TRIAL: NCT00831818
Title: Effects of Breastfeeding on Maternal Plasma Ghrelin and PYY Levels
Brief Title: Effects of Breastfeeding on Maternal Plasma Ghrelin and Peptide Tyrosine Tyrosine (PYY) Levels
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Prof. Dr. Martin Clodi, Division of Endocrinology and Metabolism, Department of Medicine III, Medical University of Vienna
Other Study IDs: Breastfeeding_01
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Breastfeeding
Keywords: breastfeeding; ghrelin; PYY; appetite-regulation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Mothers of healthy infants who breastfeed on demand
- 2: Mothers of healthy infants who do not breastfeed

SUMMARY:
Weight retention after pregnancy contributes to increasing rates of obesity. There is evidence that breastfeeding is accompanied from changes in fat mobilisation and fat mass, nevertheless there are no data on the effects of breastfeeding on appetite-regulation. This study aims to investigate the direct effect of breastfeeding on the systemic levels of appetite-regulating hormones: ghrelin and PYY. Blood samples will be obtained at five time points (before, during and after breastfeeding) in ten mothers of healthy infants who breastfeed on demand and in ten mothers of healthy infants who do not breastfeed. All mothers will be fasting since 4 hours. The results will bring information on a possible direct effect of breastfeeding on appetite-regulatory hormones.

DETAILED DESCRIPTION:
The gut-brain axis is one of the main regulators of appetite (Cummings et Overduin). Responsible for this interaction are among others the appetite-controlling gut peptides: ghrelin and PYY. Ghrelin is produced primarily in the endocrine cells of the oxyntic mucosa of the gastric fundus and was originally described as a potent endogenous GH stimulating factor (Kojima et al, Date et al). It induces short-term food intake and long-term adiposity by acting at the hypothalamus (Tschop et al, Nakazato et al). Ghrelin is highly conserved throughout the evolution and responsible for many central and peripheral endocrine and non-endocrine effects (van der Lely et al, Ghigo et al). Peptide YY or PYY is mainly produced in the terminal ileum and colon and characterized as an agent inhibiting gastrointestinal motility and appetite PYY(3-36) has been shown only recently in humans (Lundberg et al, Batterham et al. 2002). Upon infusion of PYY(3-36) subsequent food consumption was reduced in both lean and obese subjects (Batterham et al. 2003).

While the physiological and pathological control of appetite has attracted much attention in these times of increasing prevalence of obesity, nothing is known on the regulation of gut peptides during breastfeeding. Concerns that long-term weight retention after pregnancy contributes to increasing rates of obesity underscore the importance of understanding postpartum energy utilization (Mokdad et al). The 6 months following delivery of the baby are associated with a significant decrease of maternal fat mass. Fat mobilisation appears to be physiologic and gradual, even when food is readily available. Trunk fat and thigh fat are the primary energy depots mobilized to support lactation (Butte et Hopkinson). Several studies have revealed that breastfeeding facilitates post-partum weight loss (8,10). Nevertheless, it was shown that lactating women loose central and peripheral fat less rapidly then nonlactating women (Wosje et Kalkwarf). Prolonged breastfeeding has been shown to reduce the risk of developing obesity in the offspring (Cripps et al), and ghrelin has been suggested as a hormonal link between the duration of breastfeeding and body weight development (Fak et al).

The endocrinology of lactating women consists in increased amounts of prolactin and oxytocin, needed for milk production and release respectively. Very little is known on the relationship between these hormones and the appetite-modulating gut peptides. Intravenous ghrelin activates the hypothalamic-hypophysis-adrenal axis in humans and also increases prolactin release in healthy humans (Aimaretti et al). Intraventricular ghrelin administration increases intrahypothalamic oxytocin production in rats (Olszewski et al).

We recently found that continuous intravenous injection of Oxytocin decreases plasma ghrelin concentrations in healthy men (own recent and not yet published data). It is thought that increased circulating Prolactin stimulates appetite in lactating women, but there are no data on the effects of Prolactin on appetite-modulating gut hormones (Grattan). With the proposed study we aim to check the relevance of these findings in normal physiology and to study the breastfeeding-induced changes in circulating ghrelin and PYY concentrations in lactating mothers.

Setting Clinical Trial Unit of the Division of Endocrinology and Metabolism, Department of Internal Medicine III, AKH, Waehringer Gürtel 18-20, A-1090, Vienna.

Study Subjects Study group: Ten mothers of healthy infants who breastfeed on demand. Control group: Ten mothers of healthy infants who do not breastfeed.

Study Protocol

Breastfeeding group:

The study will start at ca. 10h00-12h00 and the women will be fasting since ca. 4 hours. There will be no restriction of water-intake before and throughout the study. An intravenous cannula will be inserted in the antecubital vein of one arm for blood withdrawal. The arm not needed for carrying the baby during breastfeeding will be used (e.g. if the baby is due to drink on the right breast, the intravenous cannula will be put on the left arm, und vice versa). In any case, a support cushion will be used for breastfeeding. The subjects will rest for ca. 30 minutes. Then, a basal blood withdrawal will be performed.

When the mother decides to breastfeed the baby on demand, blood will be withdrawn immediately before breastfeeding (time 0) and then at time points 15, 30 and 60 minutes. The duration of breastfeeding will be noted. 9 ml blood will be withdrawn in an EDTA-containing vacutainer at each timepoint (total 45 ml during the whole study). Ca 100µl will be separated into a cap for the online measuring of glucose, while the rest will be immediately cooled on ice and centrifuged within 30 minutes. Plasma will be aliquoted in 3 cryotubes, 2 of which will be frozen in -80°C and the third in -20°C.

Control Group:

The study will start at ca. 10h00-12h00 and the women will be fasting since ca. 4 hours. There will be no restriction of water-intake before and throughout the study. An intravenous cannula will be inserted in the antecubital vein of one arm for blood withdrawal. The subjects will rest for ca. 30 minutes. Then, a basal blood withdrawal will be performed, thereafter 4 times halfhourly.

Statistical analysis The sample number (10 breast-feeding and 10 not-breastfeeding mothers) can detect with 80% power a difference of 18% between ghrelin values after breastfeeding (α=0.05, β=0.2). Statistics will be performed using the SPSS release 12.0.1 software. Changes in hormone concentrations will be compared with repeated measures ANOVA. A possible association between parameters will be tested using linear regression analysis.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* healthy mothers (with normal BMI) fully breastfeeding their infants (aged 3 to 6 months) on demand
* past normal pregnancy

Group 2:

* healthy mothers (with normal BMI) that do not breastfeed their infants (aged 3 to 6 months)
* past normal pregnancy

Exclusion Criteria (for both groups):

* current endocrine and metabolic disease of the mother
* cardiocirculatory, kidney or liver disease of the mother
* infants having growth problems or any other current disease

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Mothers of healthy infants (babies aged 3-6 months).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
ghrelin, PYY | 60 minutes

SECONDARY OUTCOMES:
insulin, C-peptide, oxytocin, prolactin | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Martin Clodi, MD, Principal Investigator — Division of Endocrinology and Metabolism, Medical University of Vienna; Anton Luger, MD, Study Chair — Division of Endocrinology and Metabolism, Medical University of Vienna
Locations (1):
- AKH, Medical University of Vienna, Vienna, Austria